CLINICAL TRIAL: NCT00307658
Title: Intravenous Immunoglobulin After Relapse in Vasculitis (Microscopic Polyangiitis, Wegener's Granulomatosis and SHURG-STRAUSS Syndrome) During and After Corticosteroids and Immunosuppressant Therapies a Multicenter Prospective Trial
Brief Title: Intravenous Immunoglobulin After Relapse in Vasculitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P991006
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2006-05-22 (Estimated); Status verified 2003-04

CONDITIONS: ANCA + Vasculitides Relapsing Either Under Corticosteroid; and Immunosuppressant Therapies or After One Year; Post Treatment.
Keywords: ANCA associated Vasculitides; Relapse; intravenous Immunoglobulins; Corticosteroid; Immunosuppressant
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Recurrence | interventions — Immunoglobulins, Intravenous

INTERVENTIONS:
Drug: Intravenous immunoglobulins (human immunoglobulins G)

SUMMARY:
The aim of this study is to study the efficacy of intravenous immunoglobulins for inducing remission in patients relapsing of systemic vasculitides.

DETAILED DESCRIPTION:
The aim of this study will assess the effects of intravenous immunoglobulin in ANCA+ vasculitides (Microscopic Polyangiitis, Wegener's granulomatosis and Churg-Strauss syndrome) who relapse under corticosteroid and immunosuppressant therapies or after one year post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Wegener's granulomatosis, Microscopic polyangiitis and Churg-Strauss syndrome (satisfying ACR or chapel Hill classification) relapsing either under corticosteroid and immunosuppressant therapies or after one year post treatment
* Age > 18 years old
* Written informed consent

Exclusion Criteria:

* Systemic vasculitides not previously treated with corticosteroid and immunosuppressant(s)
* Systemic vasculitides treated with corticosteroids and immunosuppressant therapies, but with treatment cessation more than 12 months ago
* Polyarteritis nodosa
* Absence of poor prognosis criteria (according to FFS)
* Nephritis ± renal impairment
* Cancer or malignancy
* Psychiatric disease, lack of compliance
* Age under 18 years old
* Lack of written informed consent
* Other vasculitides (post viral infection and skin localisation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-03; Study Completion 2006-07

PRIMARY OUTCOMES:
the remission rate after 9 months of therapy with intravenous immunoglobulins,
in relapsing patients with ANCA+ vasculitides (Microscopic Polyangiitis, Wegener's granulomatosis and Churg-Strauss syndrome)
during 6 months, after relapse

SECONDARY OUTCOMES:
Safety, i.e. side-effects classified according to the WHO guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Loïc GUILLEVIN, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hopital Cochin, Paris
  - Hôpital COCHIN, Paris

REFERENCES:
- [Derived] Martinez V, Cohen P, Pagnoux C, Vinzio S, Mahr A, Mouthon L, Sailler L, Delaunay C, Sadoun A, Guillevin L; French Vasculitis Study Group. Intravenous immunoglobulins for relapses of systemic vasculitides associated with antineutrophil cytoplasmic autoantibodies: results of a multicenter, prospective, open-label study of twenty-two patients. Arthritis Rheum. 2008 Jan;58(1):308-17. doi: 10.1002/art.23147. PMID 18163506